CLINICAL TRIAL: NCT01581710
Title: A Double-blind, Randomized, Cross-over Design Study to Compare the Lung Function Measure of Montelukast Versus Placebo in Children With Mild Persistent Asthma
Brief Title: Response of FeNO, Small Airway Dysfunction and Lung Heterogeneity to 2-week Montelukast Treatment in Asthmatic Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHA University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Man Yong Han, Professor, CHA University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHA-121
Record Dates: First submitted 2012-04-13; First posted 2012-04-20 (Estimated); Results first posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Mild Persistent Asthma
Keywords: Leukotriene Antagonists; Bronchodilator response
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- montelukast to placebo (Active Comparator): 14 days
  Interventions: Drug: Montelukast to placebo
- Washout (No Intervention): 14 days
- Placebo to montelukast (Active Comparator): 14 days
  Interventions: Drug: Placebo to montelukast

INTERVENTIONS:
Drug: Montelukast to placebo — Subjects will receive montelukast (4 mg or 5 mg) Each treatment period consists of 2 weeks
  Other Names: SINGULAIR 4mg or 5mg
  Arms: montelukast to placebo
Drug: Placebo to montelukast — Subjects will receive matching placebo. Each treatment period consists of 2 weeks
  Other Names: SINGULAIR 4mg or 5mg matching placebo
  Arms: Placebo to montelukast

SUMMARY:
This study aims to identify markers to prove rapid improvement of lung function, airway inflammation and bronchodilator response after 2-week LTRA administration.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, cross-over study with a washout period of at least one week between each study period.

After an initial screening visit, subjects entered a screening period of one to two weeks to ensure clinical stability without medication, which means absence of daily asthma symptoms. Eligible subjects were randomized into either the treatment portion of the trial, in which subjects received montelukast (4 mg or 5 mg) or matching placebo monotherapy in a randomized manner. During each treatment period, which lasted 2 weeks, the study medication was administered between 8:00 and 9:00 A.M. Short acting bronchodilator (for severe symptoms) was permitted during the study period but was withheld 24 hours prior to bronchodilator challenge test.

Inclusion criteria will be mild persistent asthma children old enough to cooperate on performing pulmonary function testing, children with no respiratory symptoms 4 weeks prior to the beginning of the study. Exclusion criteria will be the following: respiratory symptoms including cough, wheezing, dyspnea, or shortness of breath, presence of acute or chronic upper respiratory infections, anatomical nasal disorders (ex, nasal polyps, septum deviation, etc.), previous or current specific immunotherapy, use of systemic corticosteroids, or admission or visit of the emergency department during the previous 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with mild persistent asthma patients based on the GINA guidelines
* children old enough to cooperate in performing pulmonary function testing
* legal guardians who sufficiently listen to the purpose and voluntarily agree with the participation to sign a written consent approved by IRB
* children with no respiratory symptoms 4 weeks prior to the beginning of the study
* children without chronic respiratory symptoms.

Exclusion Criteria:

* presence of acute or chronic upper respiratory infections, anatomical nasal disorders (ex, nasal polyps, septum deviation, etc.), previous or current specific immunotherapy.
* use of systemic corticosteroids in past 4 weeks.
* admission or visit of the emergency department in past 4 weeks.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Man Yong Han, Principal Investigator — specify Unaffiliated

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (14days)
Arm/Group | Montelukast to Placebo | Placebo to Montelukast
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: Washout Period (14days)
Arm/Group | Montelukast to Placebo | Placebo to Montelukast
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0
Period: Second Intervention (14days)
Arm/Group | Montelukast to Placebo | Placebo to Montelukast
Started | 18 | 14
Completed | 18 | 12
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Measure Analysis Population Description: two participants did not complete the second set test due to symptom aggravation
Groups:
- Subjects: All subjects
Arm/Group | Subjects
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.41 (0.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Lung function (Forced Expiratory Volume 1, predicted %) [Mean (Standard Deviation); unit: %] | 92.9 (4.4)
Lung function (Forced Expiratory Volume 1/Forced Vital Capacity, predicted %) [Mean (Standard Deviation); unit: %] | 86.1 (2.7)
oscillometric lung function (Resistance at 5Hz, z-score) [Mean (Standard Deviation); unit: z-score] | 0.36 (0.25)
oscillometric lung fuction(Reactance at 5Hz, z-score) [Mean (Standard Deviation); unit: z-score] | -1.14 (0.55)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Lung Function of Rrs 5 With IOS Before the Bronchodilator (Pre-Rrs5)
Description: Pre Rrs 5: Resistance at 5Hz before the administration of bronchodilator
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Groups:
- Baseline Lung Function: Before placebo or montelukast administration
- 2 Weeks After Placebo Administration: Subjects will receive placebo. Each treatment period consists of 2 weeks
- 2 Weeks After Montelukast Administration: Subjects will receive montelukast (4mg or 5mg) Each treatment period consists of 2 weeks
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 32 | 30 | 32
kPa/L/s | 0.73 (0.15) | 0.74 (0.20) | 0.73 (0.15)

2. Primary Outcome: Baseline Lung Function of Xrs5 With IOS Before the Bronchodilator (Pre-Xrs 5)
Description: Pre Xrs 5: Reactance at 5Hz before the administration of bronchodilator
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 32 | 30 | 32
kPa/L/s | -0.34 (0.11) | -0.36 (0.15) | -0.34 (0.10)

3. Primary Outcome: Baseline Lung Function of Rrs10 With IOS Before the Bronchodilator
Description: Pre Rrs10: Resistance at 10Hz before the administration of bronchodilator
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 32 | 30 | 32
kPa/L/s | 0.57 (0.11) | 0.55 (0.15) | 0.55 (0.12)

4. Primary Outcome: Baseline Lung Function of Xrs10 With IOS Before the Bronchodilator (Pre-Xrs10)
Description: Pre Xrs 10: Reactance at 10Hz before the administration of bronchodilator
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 32 | 30 | 32
kPa/L/s | -0.15 (0.22) | -0.20 (0.10) | -0.19 (0.07)

5. Primary Outcome: Baseline Lung Function of FEV1 Before the Bronchodilator
Description: baseline lung function in forced expiratory volume in 1 second before the administration of bronchodilator
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 32 | 30 | 32
L/s | 1.28 (0.41) | 1.25 (0.47) | 1.28 (0.46)

6. Primary Outcome: Baseline Lung Function of FEV1/FVC Before the Bronchodilator
Description: baseline lung function in forced expiratory volume in 1 second/forced vital capacity before the administration of bronchodilator
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: none (ratio)
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 32 | 30 | 32
none (ratio) | 83.55 (16.33) | 83.04 (1.22) | 85.93 (8.06)

7. Primary Outcome: Baseline Lung Function in MMEF
Description: Baseline lung function in maximal mid-expiratory flow before the administration of bronchodilator
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 32 | 30 | 32
L/s | 1.40 (0.54) | 1.38 (0.59) | 1.46 (0.50)

8. Secondary Outcome: Relative Change (%) of FEV1 After the Bronchodilator
Description: Relative change in percentage of FEV1 after the bronchodilator, 2weeks after placebo and montelukast administration Relative change (%) in FEV1 = (((FEV1 post-bronchodilator)-(FEV1 pre-bronchodilator))/baseline FEV1) x 100
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: % (relative change)
Arm/Group | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Number analyzed (Participants) | 30 | 32
% (relative change) | 9.68 (13.31) | 5.65 (10.34)

ADVERSE EVENTS:
Arm/Group | Baseline Lung Function | 2 Weeks After Placebo Administration | 2 Weeks After Montelukast Administration
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 7/30 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline Lung Function (N=32) | 2 Weeks After Placebo Administration (N=30) | 2 Weeks After Montelukast Administration (N=32)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No